CLINICAL TRIAL: NCT02583373
Title: Randomised, Multicentre, Double-blind, Placebo-controlled Study to Assess the Safety, Efficacy and Pharmacodynamics After the Intravenous Administration of CAL02 in Severe Community-acquired Pneumonia Due to Streptococcus Pneumoniae
Brief Title: Safety, Tolerability, Efficacy and Pharmacodynamics of CAL02 in Severe Pneumonia Caused by Streptococcus Pneumoniae
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combioxin SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAL02-001
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia; Pneumococcal Infections
Keywords: Pneumonia; Streptococcus pneumoniae; Pneumolysin
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CAL02 Low-dose (Active Comparator): Liposomal formulation
  Interventions: Drug: CAL02 Low-dose
- CAL02 High-dose (Active Comparator): Liposomal formulation
  Interventions: Drug: CAL02 High-dose
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAL02 Low-dose — Two doses of CAL02 (low-dose) administered 2 times (24 hours apart) as i.v. infusion
  Other Names: CAL02 LD
  Arms: CAL02 Low-dose
Drug: CAL02 High-dose — Two doses of CAL02 (high-dose) administered 2 times (24 hours apart) as i.v. infusion
  Other Names: CAL02 HD
  Arms: CAL02 High-dose
Drug: Placebo — Placebo administered administered 2 times (24 hours apart) as i.v. infusion
  Other Names: Placebo CAL02
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the safety, tolerability, clinical and microbiological efficacy and pharmacodynamics of patients who have severe pneumonia caused by Streptococcus pneumoniae after the intravenous administration of CAL02 in addition of standard of care antibiotic treatment.

DETAILED DESCRIPTION:
Streptococcus pneumoniae is the most frequently identified pathogen of community-acquired bacterial pneumonia and its severe forms are associated with high morbidity and mortality, despite pneumococcal vaccines and medical treatment (antibiotic therapy, alone or in combination). Bacterial toxins, such as the pore-forming toxin (PFT) pneumolysin (from Streptococcus pneumoniae), are involved in the development of invasive disease and play a key role in severe and fatal complications. CAL02 offers a novel therapeutic approach by neutralising bacterial toxins, such as pneumolysin, which recognise specific microdomains on host cell membranes, called lipid rafts.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients ≥ 18 years and ≤ 80 years of age
* Body weight 40-140 kg
* Severe pneumonia caused by Streptococcus pneumoniae managed in an ICU
* CURB-65 score ≥ 3 in patients aged > 65 and CURB-65 ≥ 2 in patients aged < 65
* Streptococcus pneumoniae identification with the urine antigen test or any other proven documented identification method
* Written informed consent provided by the patient, the relatives or the designated trusted person and/or according to local guidelines

Exclusion Criteria:

* Patients with hospital-acquired-, health care-acquired- or ventilator- associated-pneumonia
* More than (i) 12 hours since diagnosis of severe CAPP and (ii) 24 hours or 60 hours since antibiotic treatment IV or per os, respectively, unless documented not to be active against S. pneumoniae, will have elapsed at the time of IMP administration
* APACHE II score > 30 points
* SOFA score > 12 points
* Inability to maintain a mean arterial pressure ≥ 50 mm Hg
* Known hypersensitivity to liposomal formulations
* Patients with severe neutropenia or lymphoma or current or anticipated chemotherapy
* End-stage neuromuscular disorders
* Patients who have long-term tracheostomy
* Current or recent participation in an investigational study
* Presence of other pneumococcal site infection
* Patients with known acquired immune deficiency syndrome (AIDS) with CD4 count < 200 cells/mL
* Patients with known post-obstructive pneumonia (active primary lung cancer or another malignancy metastatic to the lungs)
* Patients with cystic fibrosis, Pneumocystis jiroveci pneumonia, or active tuberculosis
* Patients receiving immunosuppressant therapy
* Patients with a known liver function deficiency
* Splenectomised patients
* Patients who have experienced an allergic reaction to eggs
* Moribund clinical condition
* Nursing and pregnant women
* Women of child bearing potential not using an effective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Frequency, severity and characteristics of adverse events after two iv. administrations of CAL02. | 29 days
  To determine the safety profile of CAL02

SECONDARY OUTCOMES:
Clinical efficacy: cure. | 29 days.
  Complete resolution of signs and symptoms of pneumonia
Pharmacodynamic effects. | 29 days.
  Measuring biomarkers (CRP/PCT).
Microbiological efficacy. | 29 days.
  Eradication: baseline isolate not present in repeat culture from original infection site
Survival. | 29 days
  Assessment of 28 days all cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: BRUNO FRANCOIS, MD, Principal Investigator — Centre Hospitalier Universitaire de Limoges CHU Dupuytren 2 Avenue Martin Luther King 87042 Limoges Cedex, France
Locations (10):
- Belgium (3):
  - St Luc University Hospital, Brussels
  - University Hospital Brussels, Brussels
  - Clinique St Pierre, Ottignies
- France (7):
  - CHU Jean Minjoz, Besançon
  - CHD Les Oudairies, La Roche-sur-Yon
  - Hôpital Mignot, Le Chesnay
  - CHU Dupuytren, Limoges
  - Centre Hospitalier Régional d'ORLEANS, Orléans
  - CH Yves Le Foll, Saint-Brieuc
  - CHRU de Tours, Tours

REFERENCES:
- [Derived] Laterre PF, Colin G, Dequin PF, Dugernier T, Boulain T, Azeredo da Silveira S, Lajaunias F, Perez A, Francois B. CAL02, a novel antitoxin liposomal agent, in severe pneumococcal pneumonia: a first-in-human, double-blind, placebo-controlled, randomised trial. Lancet Infect Dis. 2019 Jun;19(6):620-630. doi: 10.1016/S1473-3099(18)30805-3. Epub 2019 May 2. PMID 31056427